CLINICAL TRIAL: NCT07319988
Title: A Randomized Controlled Trial Investigating the Effect of Extracorporeal Shock Wave Therapy With Core Stability Exercises for Treatment of Chronic Non-Specific Back Pain in Jordanian University Students
Brief Title: Effect of Shock Wave Therapy With Core Stability Exercises for Treatment of Chronic Non-Specific Back Pain
Acronym: ESW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New Ismailia National University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel Moeim Abo EL Ros, Assistant Professor of Pediatric Physical Therapy, New Ismailia National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB # 4/12/2024- 2025
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Back Pain
Keywords: Shock Wave; Core stability exercises; chronic non- specific back pain
MeSH Terms: conditions — Back Pain | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): will be subjected to extracorporeal shock wave therapy in addition to core stabilization exercise
  Interventions: Device: Extracorporeal Shock wave therapy
- control group (Sham Comparator): Control group will be assigned core stabilization exercises, and therapeutic ultrasound
  Interventions: Device: Extracorporeal Shock wave therapy

INTERVENTIONS:
Device: Extracorporeal Shock wave therapy — treatment of chronic non-specific back pain by shock wave therapy combined with core stabilization exercises
  Other Names: core stabilization exercise s

SUMMARY:
To investigate the Effect of Combined Extracorporeal Shock Wave with core stability Exercise for the Treatment of Chronic Non-Specific Back Pain in Jordanian University Students

DETAILED DESCRIPTION:
Chronic non-specific back pain (CNSLBP) is a prevalent condition with multifactorial causes, often linked to muscular weakness, poor postural control, and soft tissue dysfunction. Extracorporeal Shock Wave Therapy (ESWT) and core stabilization exercises (CSEs) have emerged as effective, complementary, and non-invasive treatment modalities for managing this condition.

ESWT works by delivering high-energy acoustic waves to affected tissues, stimulating biological responses such as neovascularization, collagen synthesis, and reduction of inflammation and pain mediators. These effects help improve tissue healing, decrease muscle tension, and enhance local blood flow, ultimately reducing pain intensity and improving mobility.

On the other hand, CSEs target the deep stabilizing muscles of the spine-particularly the transversus abdominis, multifidus, and pelvic floor muscles-to restore spinal stability and improve posture, balance, and functional movement. Regular performance of these exercises strengthens the core, reduces mechanical stress on the lumbar structures, and prevents pain recurrence.

When combined, ESWT and CSEs provide synergistic benefits: ESWT offers rapid pain relief and tissue recovery, facilitating better participation in exercise programs, while CSEs ensure long-term spinal stability and functional improvement. Together, they form a comprehensive and evidence-based approach to reducing pain, enhancing physical function, and improving quality of life in individuals with chronic non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* chronic non- specific back pain for more than 3 months
* teaching hours from 4 to 6 hours, 4 days per week\
* female sufferers
* Body Mass Index 20 - 22

Exclusion Criteria:

* No History of previous back surgeries
* no history of discogenic lesion
* overweight

Ages: 16 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — female
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
back pain | 12 weeks
  Measurement of pain intensity by visual analogue scale

SECONDARY OUTCOMES:
physical function | 12 weeks
  measuring of functional status by Oswestry Disability Questionnaire
Balance | 12 weeks
  Measurement of changes in balance using the Biodex Balance system

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AM Abo El Ros, Ph.D, Principal Investigator — Suez Canal University
Locations (2):
- Mohamed Abdel Moenem Abo El Ros, Ismailia, Egypt
- Zaytona University in Jordon, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No